CLINICAL TRIAL: NCT02555735
Title: Evaluation of Exceptional Responders With Solid Tumor Cancer
Brief Title: Exceptional Responders With Solid Tumor Cancer to Chemotherapy
Status: Enrolling by invitation | Type: Observational
Sponsor: Adera Labs, LLC (Industry)
Collaborators: The Pancreatic Cancer Treatment Center of Los Angeles (Unknown)
Responsible Party: Sponsor
Other Study IDs: ADRL-003
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor Neoplasms
Keywords: Solid Tumor cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Solid Tumor Cancer: Participants with solid tumor cancer treated with physician-choice standard of care chemotherapy.
  Interventions: Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: Standard of Care Chemotherapy — Physician's Choice Chemotherapy Treatment (non-guided)

SUMMARY:
This is an observational study enrolling patients with Solid Tumor cancers to identify genomic expression differences between exceptional responders and non-responders to standard of care chemotherapy. Data analysis of the gene expression profile of the exceptional responders compared to non-responders will define genomic patterns that may help understand their response to chemotherapy.

DETAILED DESCRIPTION:
This is an observational study of patients with solid tumor cancer to identify genomic expression differences obtained from their circulating tumor cells between exceptional responders and non-responders to standard of care chemotherapy. This study requires a 10 mL heparinized peripheral blood sample from each study participant at the time of enrollment to isolate, enrich and profile circulating tumor cells. Data analysis of the gene expression profile will define genomic patterns using Nearest Template Prediction for a predetermined panel of therapeutic agents based on standard of care. Chemotherapy selection is physician-choice. Information regarding disease progression will be gathered. Data analysis will be performed in study participants in the setting of ongoing disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of solid tumor carcinoma.
* Patient is treatment-naïve or currently receiving chemotherapy.
* ECOG performance status (any).

Exclusion Criteria:

* HIV positive on antiretroviral therapy
* Pregnant or lactating
* Prior organ allograft
* Any medical or psychiatric condition that may interfere with the ability to comply with protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with solid tumor cancers
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2015-10; Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Identify exceptional responders with cancer to standard of care chemotherapy | 9 years
  Identify responders and non-responders

SECONDARY OUTCOMES:
Correlation of genomic profiles from circulating cells with overall survival | 9 years
  Genomic expression profiles correlated with progression free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Brian McCarthy, PhD, Study Director — Adera Labs
Locations (1):
- The Pancreatic Cancer Treatment Center of Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Yu KH, Ricigliano M, McCarthy B, Chou JF, Capanu M, Cooper B, Bartlett A, Covington C, Lowery MA, O'Reilly EM. Circulating Tumor and Invasive Cell Gene Expression Profile Predicts Treatment Response and Survival in Pancreatic Adenocarcinoma. Cancers (Basel). 2018 Nov 24;10(12):467. doi: 10.3390/cancers10120467. PMID 30477242
- [Background] Isacoff WH, Cooper B, Bartlett A, McCarthy B, Yu KH. ChemoSensitivity Assay Guided Metronomic Chemotherapy Is Safe and Effective for Treating Advanced Pancreatic Cancer. Cancers (Basel). 2022 Jun 13;14(12):2906. doi: 10.3390/cancers14122906. PMID 35740571
- [Background] Yu KH, Park J, Mittal A, Abou-Alfa GK, El Dika I, Epstein AS, Ilson DH, Kelsen DP, Ku GY, Li J, Park W, Varghese AM, Chou JF, Capanu M, Cooper B, Bartlett A, McCarthy D, Sangar V, McCarthy B, O'Reilly EM. Circulating tumor and invasive cell expression profiling predicts effective therapy in pancreatic cancer. Cancer. 2022 Aug 1;128(15):2958-2966. doi: 10.1002/cncr.34269. Epub 2022 Jun 1. PMID 35647938